CLINICAL TRIAL: NCT00594763
Title: The Risk of Venous Thrombosis in Women With Turner Syndrome
Brief Title: Venous Thrombosis in Turner Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Jens Sandahl Christiansen, Aarhus University Hospital, Aarhus, Denmark
Other Study IDs: 20050045
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Thromboembolic Disease
Keywords: Turner syndrome; Thromboembolic disease
MeSH Terms: conditions — Thromboembolism; Turner Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TS: Women with Turner syndrome

SUMMARY:
In the literature, cases of thrombosis in the venous system have been described in girls and women with Turner syndrome. By screening a group of women with Turner syndrome, the researchers wish to find out if this condition is more frequent in this patient population.

DETAILED DESCRIPTION:
In the literature cases of thrombosis in the venous system has been described in girls and women with Turner syndrome. By screening a group of women with Turner syndrome we wish to find out if this condition is more frequent in this patient population. Participants are examined with screening blood tests evaluating thromboembolic disturbances.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome verified by karyotyping
* Aged 18 or above

Exclusion Criteria:

* Malignant disease
* Treatment with anticoagulants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with Turner syndrome
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-04 (Estimated); Study Completion 2008-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Sandahl Christiansen, MD, dr.med, professor, Principal Investigator — Medical Department of Endocrinology, Aarhus University Hospital, 8000 Aarhus, Denmark
Locations (1):
- Medical Department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, Aarhus C, Denmark